CLINICAL TRIAL: NCT07172321
Title: A Phase 1, Open-Label, Randomized, 5-Period, 6-Sequence, Crossover Study to Compare the Single-Dose Pharmacokinetics of One Immediate-Release and Two Modified-Release Formulations of PF-08049820 Administered Orally to Healthy Adult Participants Under Fasted and Fed Conditions
Brief Title: A Study to Learn How Different Forms of the Study Medicine Called PF 08049820 Are Taken up Into the Bloodstream in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C6231007
Record Dates: First submitted 2025-08-28; First posted 2025-09-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: Healthy Volunteer
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Treatment A (Experimental): Participants will receive a single dose of PF-08049820 short Modified release (MR) release rate (MR1) tablets under fasted conditions.
  Interventions: Drug: PF-08049820 MR1
- Treatment B (Experimental): Participants will receive a single dose of PF-08049820 long MR release rate (MR2) tablets under fasted conditions.
  Interventions: Drug: PF-08049820 MR2
- Treatment C (Experimental): Participants will receive a single dose of PF-08049820 Immediate Release (IR) tablets under fasted conditions.
  Interventions: Drug: PF-08049820 IR
- Treatment D (Experimental): Participants will receive a single dose of PF-08049820 MR2 tablets under fed conditions.
  Interventions: Drug: PF-08049820 MR2
- Treatment E (Experimental): Participants will receive a single dose of PF-08049820 IR tablets under fed conditions.
  Interventions: Drug: PF-08049820 IR

INTERVENTIONS:
Drug: PF-08049820 MR1 — Administered orally
  Arms: Treatment A
Drug: PF-08049820 MR2 — Administered orally
  Arms: Treatment B; Treatment D
Drug: PF-08049820 IR — Administered orally
  Arms: Treatment C; Treatment E

SUMMARY:
The purpose of this study is to see how different forms of a medicine called PF-08049820 move through the body when taken by mouth. The scientists want to see:

* How well is the medicine absorbed when it's made in different ways (fast vs. slow release)
* If eating a high-fat meal changes how the medicine moves through the body The results of this study will help decide which version of the medicine is best for future studies.

This study is seeking participants who:

* are men and women who can't have children
* are 18 years or older
* weigh more than 99 pounds (45 kg)
* have a healthy body weight (not too low or too high)
* are generally healthy with no serious medical problems. People with serious health problems, recent drug use, or who had certain vaccines recently cannot join.
* are willing to follow all the study rules

Each participant will try 5 different versions of the medicine, one at a time. There will be 3 days between each dose to make sure the medicine is out of the system. The medicine will be tested in different forms:

* Immediate-release tablet (works quickly)
* Short-release tablet (works slowly)
* Long-release tablet (works even slower)

Some versions will be taken without food, and others after eating a high-fat meal. After each dose, doctors will take blood samples for up to 72 hours to see how the medicine moves through the body. The whole study will take about 6 to 11 weeks and participants will stay overnight in the clinic for about 17 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants of non-childbearing potential ≥18 years of age
* BMI of 16-32 kg/m2; and a total body weight >45 kg (99 lbs)
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

  * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
  * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBsAb, HBcAb, or HCVAb. A positive HBsAb result and a history of Hepatitis B vaccination is allowed.
* Use of certain prescription or nonprescription drugs and dietary (e.g. grapefruit) and herbal supplements within up to 14 days or 5 half-lives, whichever is longer, prior to the first dose of study intervention.
* Recent exposure to live or attenuated vaccines within 28 days of the screening visit.
* Previous administration of an investigational product (drug or vaccine) within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Plasma Area Under the Concentration Versus Time Curve (AUC) of PF-08049820 in the fasted state | Pre-dose until 72 hours post dose
PK: Plasma Maximum Concentration (Cmax) of PF-08049820 in the fasted state | Pre-dose until 72 hours post dose

SECONDARY OUTCOMES:
PK: Plasma Area Under the Concentration Versus Time Curve (AUC) of PF-08049820 in the fed state | Pre-dose until 72 hours post dose
PK: Plasma Maximum Concentration (Cmax) of PF-08049820 in the fed state | Pre-dose until 72 hours post dose
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | First dose, up to follow up visit (28-35 days post last dose)
Number of Participants With Clinical Laboratory Abnormalities | Baseline, up to Day 16
Number of Participants With Vital Signs Abnormalities | Baseline, up to Day 16
Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings | Baseline, up to Day 16

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6231007